CLINICAL TRIAL: NCT06918184
Title: Timing of Specific Exercise Therapy After Breast Cancer Surgery: A Single-Center, Parallel-Group Randomized Controlled Trial Comparing Early (<1 Week Postoperative) Versus Delayed (3 Weeks Postoperative) Initiation for Optimized Upper Limb Function
Brief Title: Timing of Specific Exercise Therapy After Breast Cancer Surgery: Early Versus Delayed Initiation
Acronym: BEST-Timing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCExTiming2025-02
Record Dates: First submitted 2025-03-30; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible women will be randomly assigned to either the early or delayed specific exercise therapy initiation group. The interventions will be identical aside from the timing; both groups will receive supervised exercise sessions and subsequent home maintenance.
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the intervention timing, participants, care providers, and investigators are unblinded; however, those assessing the primary and secondary outcomes will be blinded to treatment group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Initiation of Specific Exercise Therapy (Experimental): In this group, participants will initiate specific exercise therapy within the first postoperative week. They will receive 40-minute supervised sessions twice weekly for 8 weeks, with a transition to a prescribed home-based maintenance program for an additional 4 months.
  Interventions: Behavioral: Specific Exercise Therapy
- Delayed Initiation of Specific Exercise Therapy (Experimental): Participants in this group will begin the same specific exercise therapy protocol at 3 weeks postoperative. Otherwise, the intervention is identical to that provided to the Early Therapy group.
  Interventions: Behavioral: Specific Exercise Therapy

INTERVENTIONS:
Behavioral: Specific Exercise Therapy — The exercise protocol includes mobilisation and stretching with 40-minute sessions twice weekly for 8 weeks post-initiation, transitioning to a home-based maintenance phase for 4 months. All sessions will be supervised by certified physiotherapists.

SUMMARY:
This single-center, parallel-group randomized controlled trial (RCT) will compare two timings for initiating specific exercise therapy after breast cancer surgery. The study tests whether early initiation (within the first postoperative week) versus delayed initiation (at 3 weeks postoperative) results in superior upper limb function at 6 months as measured by the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire. Secondary outcomes include pain intensity (Visual Analog Scale, VAS) and wound-related complications such as drainage time and hematoma incidence.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-65 years.
* Scheduled to undergo breast cancer surgery with axillary node dissection.
* At risk for upper limb morbidity based on preoperative assessment.
* Able to provide informed consent and complete study questionnaires.
* Willing and able to attend scheduled physiotherapy sessions and follow-up evaluations.

Exclusion Criteria:

* Diagnosis of recurrent or metastatic breast cancer.
* Concurrent participation in another rehabilitation intervention or clinical trial.
* Severe comorbidities (e.g., uncontrolled cardiovascular disease, severe orthopedic conditions) that preclude safe participation.
* History of previous shoulder surgery or chronic upper extremity musculoskeletal disorders unrelated to breast cancer treatment.
* Inability to understand or complete study materials in English.
* Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Upper Limb Function (DASH Questionnaire) | Assessed preoperatively (baseline) and at 6 months postoperative.
  The Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire is a validated measure of upper limb function. The questionnaire is scored on a continuous scale ranging from 0 to 100, where 0 indicates no disability and 100 represents the most severe disability. Lower scores indicate better upper limb function.

SECONDARY OUTCOMES:
Pain Intensity (Visual Analog Scale - VAS) | Assessed at baseline and at 1, 3, and 6 months postoperative.
  A 0-100 VAS will measure patient-reported pain levels, where 0 signifies no pain and 100 the worst pain imaginable.
Wound-Related Complications - Drainage Time (Days) | Monitored during the immediate postoperative period up to 3 months.
  The duration of wound drainage will be recorded in days. Longer drainage time may indicate wound complications.
Wound-Related Complications - Incidence of Hematoma | Monitored during the immediate postoperative period up to 3 months.
  The occurrence of hematoma will be documented as a binary outcome (presence or absence) for each patient. The incidence will be calculated as the proportion of patients developing hematoma during the monitoring period.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Al Hayah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No